CLINICAL TRIAL: NCT03062774
Title: The Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Study of Continuous Multiple Dose PB-119 Injection in Health Volunteers
Brief Title: Continuous Multiple Dose PB-119 Injection in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICP-2014-07
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PB-119 (Experimental): intervention: PB-119 injection
  Interventions: Biological: PB-119 injection

INTERVENTIONS:
Biological: PB-119 injection

SUMMARY:
This is an open label, multiple dose study, pharmacokinetic and pharmacodynamics studies will be performed at the same time with tolerability study. Three dose arms are designed, 12 subjects will be enrolled in each arm, will equal number of males and females.

DETAILED DESCRIPTION:
Pharmacokinetic and pharmacodynamics studies were performed in parallel with PB-119 25μg、50μg、and 100μg dose escalation tolerability study, plasma samples were collected to determine drug concentration and pharmacodynamics parameters. The study duration of each arm was 8 weeks, study medication was given about 8:00 a.m. on day 1 of each week, totally 6 times, and subject was followed until 15 days after last dose (50 days of study) and then study can be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects between the ages of 18~45 years at screening;
2. Weight: female weight of ≥45 kg, male weight of ≥50 kg, subject body mass index (BMI) between 19~30 kg/m2 (inclusive);
3. Pretrial physical examination, blood routine test, urine routine test, liver and kidney function and related laboratory examination results are normal or mildly abnormal but determined by investigator as no clinical significance;
4. Fasting blood glucose (FPG) results of ≤ 6.0mmol / L;
5. Subjects must be consented before study, and willing to sign the written informed consent;
6. Subjects are able to well communicated with investigators, comply with study procedure and complete study.

Exclusion Criteria:

1. Specific allergy to investigational drug or any ingredients (citric acid, mannitol, m-cresol);
2. Have clinical significant major disease or major surgery within 4 weeks before study initiation.
3. Have any clinical significant major disease history or medical history of circulatory system, endocrine system, nervous system disease or hematology, immunology, psychiatric diseases and metabolic disorders etc.
4. Have history of gastrointestinal, liver and kidney disease (for example: have liver, kidney or gastrointestinal partial resection surgery );
5. Have fever before 3 days of screening;
6. The screening laboratory tests (blood routine test, urine routine test, blood biochemical tests, etc.) were determined by investigator as abnormal with clinical significance within 2 weeks before study initiation;
7. Pretrial electrocardiogram and vital signs were determined as clinically significant abnormal by investigator (systolic blood pressure <90 mmHg or ≥ 140 mmHg, diastolic blood pressure <60 mmHg or ≥ 90 mmHg; heart rate <50 bpm or> 100 bpm);
8. Positive of HIV, hepatitis B surface antigen, hepatitis C, Treponema pallidum antibody test；
9. Alcoholic or frequent drinkers within 6 months before trial, ie more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol contented spirit or 150 mL of wine);
10. Heavily smoker or more than 5 cigarettes per day within 3 months before trial, or any tobacco product used during trial;
11. Drug abusers or those who have used soft drugs (e.g. marijuana) 3 months prior to the trial or those who took hard drugs (e.g. cocaine, phencyclidine, etc.) one year before and during the trial;
12. Allergy to any food or has special requirement to food, not be able to comply to unify diet;
13. Excessive consumption of tea, coffee and / or caffeinated beverages (8 cups or more) per day;
14. Take any medications that may affect test results, such as antibiotics, non-steroidal anti-inflammatory drugs, antacids containing aluminum or magnesium, diuretics, anticoagulants, central nervous system inhibitors, and any drug that may possibly affect the absorption of the drug within 2 weeks before screening;
15. Take any clinical trial investigational medication or participate any drug clinical trial within 3 months before trial;
16. Blood donation up to or more than 360ml within 3 months before screening;
17. Female subjects who plan pregnancy or male subjects who's spouse plan to be pregnant within 6 months;
18. Female subjects who take oral contraceptive within 30 days before and during trial;
19. Female who received long-acting estrogen or progestin injections or implants within 6 months before and during the trial;
20. Female of childbearing potential had non-protective sexual intercourse with partner within 14 days before and during trial;
21. Female who is pregnant or lactating;
22. Subject who cannot complete study due to other reason or determined by investigators as inappropriate to participate this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Change from Baseline lab value at 50 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Determine PB-119 blood concentration | Day1-8, Day 15, Day 22, Day 29, Day 36-42, Day 46,Day 50, Day 54 and Day 58
  Number of PB-119 blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yuan LV, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui H, Zhao CY, Lv Y, Wei MJ, Zhu Y, Ma XZ, Xia YH, Tian JH, Ma Y, Liu Y, Zhang P, Xu M. Safety, Pharmacokinetics and Pharmacodynamics of Multiple Escalating Doses of PEGylated Exenatide (PB-119) in Healthy Volunteers. Eur J Drug Metab Pharmacokinet. 2021 Mar;46(2):265-275. doi: 10.1007/s13318-020-00665-x. Epub 2021 Feb 12. PMID 33576936